CLINICAL TRIAL: NCT04674579
Title: The Added Value of Automatic Segmentation of Cerebral Gliomas in Multi-Sequence Magnetic Resonance Imaging (MRI)
Brief Title: Automatic Segmentation MRI Cerebral Glioma
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Fatma Rabiee Ali Sedeek, assuit egypt, Assiut University
Other Study IDs: MRI cerebral glioma
Record Dates: First submitted 2020-12-14; First posted 2020-12-19 (Actual); Last update posted 2020-12-19 (Actual); Status verified 2020-12

CONDITIONS: Cerebral Glioblastoma
Keywords: MRI automatic segmentation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: MRI — magnetic resonance imaging

SUMMARY:
The aim of this study is to evaluate the role of automatic segmentation of cerebral gliomas in multi-sequence MR images using state-of-the-art methods for automatic segmentation and internal classification of brain tumors in correlation with operative findings

DETAILED DESCRIPTION:
Gliomas are the most common primary brain tumors and are classified by their histopathological appearances using the World Health Organization (WHO) system into low-grade glioma (LGG) (grades I and II) and high-grade glioma (grade III anaplastic glioma and grade IV glioblastoma.

Gliomas, particularly high-grade, exhibit irregular growth patterns infiltrating the surrounding brain and thus showing irregular boundaries that may not be clear on conventional magnetic resonance images (MRI) MR images are visually inspected by radiologists, however, visual assessment is subjective, time consuming and prone to variability due to inter-rater differences. Accurate delineation of tumor boundaries as well as assessment of tumor volume are essential for treatment planning and monitoring treatment response . However, accurate delineation of the boundaries of glioma using subjective visual assessment is often difficult due to tumor heterogeneity and complexity, overlapping signal intensity with surrounding tissues and uneven tumor growth into nearby structures .

Compared to tumor volumetry, the routine visual evaluation of tumor size is based upon simple linear measurements of the gross tumor volume. These bi-dimensional measurements are often performed on a single MRI slice without volumetric measurements. These linear measurements are user-dependent and prone to errors due to increased measurement variability, especially in irregularly shaped lesions Computer-based fully-automatic tumor segmentation methods present a possible solution to these issues. The process is based upon information extraction from structural brain MRI images using a probabilistic tissue model to define the clear tumor boundaries using different MRI pulse sequences. These methods could accurately and rapidly identify glioma from surrounding normal brain tissue, and perform tumor volumetry, while eliminating intra-observer and inter-observer variability Internal changes within glioma, such as enhancement pattern and degeneration are crucial for identification of glioma grade, planning of treatment, monitoring of disease progression and evaluating the efficacy of therapy. In the process of automatic glioma segmentation, different parts of the glioma are characterized as solid (active) tumor, necrosis and peri-tumoral edema .

Automatic segmentation methods utilize artificial intelligence and machine learning techniques for extraction of information from multi-sequence MRI including, basically, T1W, Gadolinium enhanced T1W, T2W and FLAIR sequences .

Appropriate assessment of the extent of tumor resection plays an important role in the prognosis of glioma, since maximizing the extent of resection influences survival in these patients. Complete resection of enhancing tumor, defined as the removal of the final 1-2% of the tumor, seems to provide the most benefit in terms of patient's survival . Automatic segmentation could lead to better diagnosis and proper treatment planning through accurate tumor localization and classification .

ELIGIBILITY:
Inclusion Criteria:

- Patients with cerebral gliomas identified by MRI who will be treated surgically

Exclusion Criteria:

* Previously operated or biopsied gliomas.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: The study will include 50 patients with cerebral gliomas identified by MRI A standardized multi-parametric MR protocol will be implemented for all patients. All sequences will be acquired on a 1.5T MR scanner.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2021-01-01 (Estimated); Primary Completion 2023-02 (Estimated); Study Completion 2023-04 (Estimated)

PRIMARY OUTCOMES:
evaluate the role of automatic segmentation of cerebral gliomas in multi-sequence MR images in correlation with operative findings. | baseline
  The aim of this study is to evaluate the role of automatic segmentation of cerebral gliomas in multi-sequence MR images using state-of-the-art methods for automatic segmentation and internal classification of brain tumors in correlation with operative findings.

CONTACTS AND LOCATIONS:
Overall Officials: Mostafa Mostafa, Study Director — Assiut University; Hosameldeen Metwalli, Study Director — Assiut University; Noha Attia, Study Director — Assiut University; fatma sedeek, Principal Investigator — Assiut University

REFERENCES:
- [Background] Soltaninejad M, Yang G, Lambrou T, Allinson N, Jones TL, Barrick TR, Howe FA, Ye X. Automated brain tumour detection and segmentation using superpixel-based extremely randomized trees in FLAIR MRI. Int J Comput Assist Radiol Surg. 2017 Feb;12(2):183-203. doi: 10.1007/s11548-016-1483-3. Epub 2016 Sep 20. PMID 27651330
- [Background] Wen PY, Macdonald DR, Reardon DA, Cloughesy TF, Sorensen AG, Galanis E, Degroot J, Wick W, Gilbert MR, Lassman AB, Tsien C, Mikkelsen T, Wong ET, Chamberlain MC, Stupp R, Lamborn KR, Vogelbaum MA, van den Bent MJ, Chang SM. Updated response assessment criteria for high-grade gliomas: response assessment in neuro-oncology working group. J Clin Oncol. 2010 Apr 10;28(11):1963-72. doi: 10.1200/JCO.2009.26.3541. Epub 2010 Mar 15. PMID 20231676
- [Background] Niyazi M, Brada M, Chalmers AJ, Combs SE, Erridge SC, Fiorentino A, Grosu AL, Lagerwaard FJ, Minniti G, Mirimanoff RO, Ricardi U, Short SC, Weber DC, Belka C. ESTRO-ACROP guideline "target delineation of glioblastomas". Radiother Oncol. 2016 Jan;118(1):35-42. doi: 10.1016/j.radonc.2015.12.003. Epub 2016 Jan 6. PMID 26777122
- [Background] Tabatabai G, Stupp R, van den Bent MJ, Hegi ME, Tonn JC, Wick W, Weller M. Molecular diagnostics of gliomas: the clinical perspective. Acta Neuropathol. 2010 Nov;120(5):585-92. doi: 10.1007/s00401-010-0750-6. Epub 2010 Sep 23. PMID 20862485
- [Background] Kanaly CW, Mehta AI, Ding D, Hoang JK, Kranz PG, Herndon JE 2nd, Coan A, Crocker I, Waller AF, Friedman AH, Reardon DA, Sampson JH. A novel, reproducible, and objective method for volumetric magnetic resonance imaging assessment of enhancing glioblastoma. J Neurosurg. 2014 Sep;121(3):536-42. doi: 10.3171/2014.4.JNS121952. Epub 2014 Jul 18. PMID 25036205
- [Background] Meier R, Knecht U, Loosli T, Bauer S, Slotboom J, Wiest R, Reyes M. Clinical Evaluation of a Fully-automatic Segmentation Method for Longitudinal Brain Tumor Volumetry. Sci Rep. 2016 Mar 22;6:23376. doi: 10.1038/srep23376. PMID 27001047
- [Background] Gordillo N, Montseny E, Sobrevilla P. State of the art survey on MRI brain tumor segmentation. Magn Reson Imaging. 2013 Oct;31(8):1426-38. doi: 10.1016/j.mri.2013.05.002. Epub 2013 Jun 20. PMID 23790354
- [Background] Porz N, Habegger S, Meier R, Verma R, Jilch A, Fichtner J, Knecht U, Radina C, Schucht P, Beck J, Raabe A, Slotboom J, Reyes M, Wiest R. Fully Automated Enhanced Tumor Compartmentalization: Man vs. Machine Reloaded. PLoS One. 2016 Nov 2;11(11):e0165302. doi: 10.1371/journal.pone.0165302. eCollection 2016. PMID 27806121
- [Background] Naceur MB, Saouli R, Akil M, Kachouri R. Fully Automatic Brain Tumor Segmentation using End-To-End Incremental Deep Neural Networks in MRI images. Comput Methods Programs Biomed. 2018 Nov;166:39-49. doi: 10.1016/j.cmpb.2018.09.007. Epub 2018 Sep 21. PMID 30415717